CLINICAL TRIAL: NCT00600743
Title: Effect of a CCK-1R Agonist on Food Intake in Humans
Acronym: GSK
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug expired before was completed.
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 07-101
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Bulimia
Keywords: Eating; Food Intake; Appetite
MeSH Terms: conditions — Bulimia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- 1 'Instructions to eat normally' (Placebo Comparator): 'Instructions to eat normally' Placebo 1 mg dose
  Interventions: Behavioral: Instructions to eat normally; Drug: Placebo
- 2 'Instructions to eat normally' (Active Comparator): 'Instructions to eat normally' drug 1 mg dose 'GSKI181771X (CCK-1R agonist)'
  Interventions: Drug: GSKI181771X (CCK-1R agonist); Behavioral: Instructions to eat normally
- 3 'Instructions to eat normally' (Placebo Comparator): 'Instructions to eat normally' 2 mg placebo
  Interventions: Behavioral: Instructions to eat normally; Drug: Placebo
- 4 'Instructions to eat normally' (Active Comparator): 'Instructions to eat normally' 2 mg drug 'GSKI181771X (CCK-1R agonist)'
  Interventions: Drug: GSKI181771X (CCK-1R agonist); Behavioral: Instructions to eat normally
- 5 'Instructions to eat normally' (Placebo Comparator): 'Instructions to eat normally' 4 mg placebo
  Interventions: Behavioral: Instructions to eat normally; Drug: Placebo
- 6 'Instructions to eat normally' (Active Comparator): 'Instructions to eat normally' 4 mg drug 'GSKI181771X (CCK-1R agonist)'
  Interventions: Drug: GSKI181771X (CCK-1R agonist); Behavioral: Instructions to eat normally
- 7 Instructions to binge eat (Placebo Comparator): Instructions to binge eat 4 mg placebo
  Interventions: Behavioral: Instructions to binge eat; Drug: Placebo
- 8 Instructions to binge eat (Active Comparator): Instructions to binge eat 4 mg drug 'GSKI181771X (CCK-1R agonist)'
  Interventions: Drug: GSKI181771X (CCK-1R agonist); Behavioral: Instructions to binge eat

INTERVENTIONS:
Drug: GSKI181771X (CCK-1R agonist) — Drug one trial vs placebo
  Other Names: GSKI181771X
  Arms: 2 'Instructions to eat normally'; 4 'Instructions to eat normally'; 6 'Instructions to eat normally'; 8 Instructions to binge eat
Behavioral: Instructions to binge eat — Subjects will be instructed to binge eat and will also be given either drug or placebo
  Arms: 7 Instructions to binge eat; 8 Instructions to binge eat
Behavioral: Instructions to eat normally — Subjects will be instructed to eat normally and will also be given either drug or placebo
  Arms: 1 'Instructions to eat normally'; 2 'Instructions to eat normally'; 3 'Instructions to eat normally'; 4 'Instructions to eat normally'; 5 'Instructions to eat normally'; 6 'Instructions to eat normally'
Drug: Placebo — Drug one trial vs placebo
  Arms: 1 'Instructions to eat normally'; 3 'Instructions to eat normally'; 5 'Instructions to eat normally'; 7 Instructions to binge eat

SUMMARY:
The ultimate aim of this study is to test the hypothesis that the oral cholecystokinin (CCK) agonist GSKI181771X will reduce the size of a binge meal among individuals with Bulimia Nervosa. The study will be conducted in phases. First, an effective dose for reducing food intake, when normal subjects eat normally will be attained. Next, it will be determined whether intake at this dose is reduced in control subjects instructed to eat to capacity. If the dose is still effective compared to placebo, the same dose will be tested in patients with bulimia nervosa.

DETAILED DESCRIPTION:
This study tests the hypothesis that an oral CCK antagonist GSKI181771X will reduce the size of a binge meal. It was intended to study the effects of increasing doses on antagonist on normal individuals to find an effective dose in a non-binge meal before moving to a binge meal. Once the effects of the antagonist on a binge meal were found, the compound would be used on patients with bulimia nervosa. However, the product expired and more was not available before the patients were tested. Data are presented for the normal participants who were instructed to eat normally, followed by a group that was instructed to binge eat. Comparisons were made between groups with different instructions and between binge and normal meals.

ELIGIBILITY:
Inclusion Criteria:

* Both controls and patients will be female, 18 to 45 years old, and within 80-120% of ideal body weight (Metropolitan Life Insurance, 1983). Inclusion and exclusion will be evaluated using the following guidelines:

Normal Controls:

* No current or past psychiatric illness
* No history of binge eating or vomiting
* 80-120% ideal weight
* Of non-childbearing potential (i.e. physiologically incapable of becoming pregnant or surgically sterile)
* If of childbearing potential, willing to use an acceptable method of birth-control (please see list in "Exclusion" section)

Patients with Bulimia Nervosa:

* DSM-IV (diagnostic statistical manual - American Psychiatric Association) criteria for bulimia nervosa
* Duration of illness > 1 year
* Purging after binges via self-induced vomiting

(Same as controls for remaining inclusion criteria)

Exclusion Criteria:

Normal Controls:

* Significant medical illness: CBC, Chem-1, serum electrolytes (sodium, potassium, chloride, CO2), glucose, BUN (blood urea nitrogen), creatinine, Alk Phos, ALT (SGPT), AST (SGOT), LDH, total bilirubin, total protein, albumin, globulin, A/G ratio, calcium, phosphorus, uric acid, cholesterol, triglyceride
* ALT outside of upper limit of normal: Chem-1
* History of gallstones, pancreatitis or cholecystitis
* Current medication
* Hypersensitivity to benzodiazepines (contraindication in DCSI v02, 1-March-2006)
* Drug or alcohol abuse in last 3 mts
* Pregnancy
* Unable or unwilling to use highly effective methods of contraception for the duration of the study until an insignificant amount of the investigational product remains in the subject (i.e. at least 5 terminal phase half-lives). Examples of highly effective methods of contraception are:

  * Implants of levonorgestrel, or
  * Injectable progestogen, or
  * Oral birth control pills for at least 3 monthly cycles prior to administration of study drug + continuation for 24 hrs after last dose of study drug, or
  * Double-barrier method (e.g. condom, diaphragm) with spermicide

Note-Significant medical illness is any illness requiring continued care, i.e. chronic medication. Examples include hypertension, diabetes, and systemic lupus erythematosis. Subjects with seasonal allergies or occasional urinary tract infections will be included.

Patients with Bulimia Nervosa:

* Same as controls

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry R. Kissileff, Ph.D., Principal Investigator — St. Luke's-Roosevelt Hospital Center; Jeanine Albu, MD, Study Director — St. Luke's-Roosevelt Hospital Center
Locations (1):
- St. Luke's/Roosevelt Hospital, New York, New York, United States

REFERENCES:
- See also: studies — http://www.nyorc.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment at St. Luke's Hospital from 2/22/08 through 2/19/09
Pre-assignment Details: Subject had to rate test food greater than 6 on a 9 point scale of liking and have BMI between 19 and 27
Groups:
- 1 MG CCK AGONIST NORMAL EATING: Healthy/normal control participants were given both the 1 mg oral cholecystokinin (CCK) agonist (GSKI181771X) and placebo interventions at separate times in a 2 way crossover study design. After ingesting the CCK agonist or placebo, they were instructed to eat until they felt normally full.
- 2 MG CCK AGONIST NORMAL EATING: Healthy/normal control participants were given both the 2 mg oral cholecystokinin (CCK) agonist (GSKI181771X) and placebo interventions at separate times in a 2 way crossover study design. After ingesting the CCK agonist or placebo, they were instructed to eat until they felt normally full.
- 4 MG CCK AGONIST NORMAL EATING: Healthy/normal control participants were given both the 4mg oral cholecystokinin (CCK) agonist (GSKI181771X) and placebo interventions at separate times in a 2 way crossover study design. After ingesting the CCK agonist or placebo, they were instructed to eat until they felt normally full.
- 4 MG CCK AGONIST BINGE EATING: Healthy/normal control participants were given both the 4 mg oral cholecystokinin (CCK) agonist (GSKI181771X) and placebo interventions at separate times in a 2 way crossover study design. After ingesting the CCK agonist or placebo, they were instructed to binge eat as much as they could.
Period: Overall Study
Arm/Group | 1 MG CCK AGONIST NORMAL EATING | 2 MG CCK AGONIST NORMAL EATING | 4 MG CCK AGONIST NORMAL EATING | 4 MG CCK AGONIST BINGE EATING
Started | 4 | 4 | 8 | 7
Completed | 4 | 4 | 8 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 MG CCK AGONIST NORMAL EATING | 2 MG CCK AGONIST NORMAL EATING | 4 MG CCK AGONIST NORMAL EATING | 4 MG CCK AGONIST BINGE EATING | Total
Number analyzed (Participants) | 4 | 4 | 8 | 7 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (10.96) | 26.25 (3.0) | 23.75 (10.77) | 24.00 (11.64) | 24.65 (3.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8 | 7 | 23
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8 | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Food Intake for 4 mg Dose of CCK Agonist vs Placebo Meal Conditions
Description: Food Intake at 25-30 min after having drug or placebo under normal and binge eating instructions
Time Frame: 25-30 min after taking drug
Population: Subjects had to complete all trials of the protocol successfully
Measure: Mean (Standard Error); unit: grams
Groups:
- Binge_4mg Drug: Non-bulimic controls Instruction to binge eat (7 subjects) drug
- Normal_1mg Drug: Eat normally 1 mg dose drug
- Normal_2mg Drug: Eat normally 2 mg dose drug
- Normal_4mg Drug: Eat normally 4 mg dose drug
- Binge - 4mg Placebo: Non-bulimic controls instruction to binge eat - placebo
- Normal 1 mg Dose Placebo: Eat normally 1 mg dose placebo
- Normal_2 mg Dose Placebo: Eat normally 2 mg dose placebo
- Normal_4 mg Dose Placebo: Eat normally 4 mg dose placebo
Arm/Group | Binge_4mg Drug | Normal_1mg Drug | Normal_2mg Drug | Normal_4mg Drug | Binge - 4mg Placebo | Normal 1 mg Dose Placebo | Normal_2 mg Dose Placebo | Normal_4 mg Dose Placebo
Number analyzed (Participants) | 7 | 4 | 4 | 8 | 7 | 4 | 4 | 8
grams | 385.69 (29.35) | 447.7 (38.64) | 489.63 (45.54) | 293.79 (65.58) | 532.87 (53.4) | 468.73 (74) | 442.43 (61.79) | 421.98 (69.26)
Statistical Analysis 1: Comparison: Normal_4mg Drug vs Normal_4 mg Dose Placebo; Repeated measures ANOVA; Test type: Superiority or Other; p = 0.007, t-test, 2 sided — t test following ANOVA for difference between drug and placebo - There were 3 doses, and the value reported is for the highest and only effective dose; The overall error term was used to compare differences between placebo and drug; Mean Difference (Final Values) = 128.2, Standard Error of Mean 41.4

2. Secondary Outcome: Fullness Rating
Description: rating of "How full do you feel" by marking the feeling on a 150 mm line anchored at one end from 0 (not at all) to 150 (most imaginable).
Time Frame: 25-30 min after taking drug
Measure: Mean (Standard Error); unit: mm
Groups:
- Binge_4mg d: Binge_4mg drug
- Normal_1mg d: Normal_1mg drug
- Normal_2mg d: Normal_2mg drug
- Normal_4mg d: Normal_4mg drug
- Binge - 4mg Plc: binge - 4mg placebo
- Normal 1 mg Placebo: Normal 1 mg dose placebo
- Normal 2mg_placebo: Normal 2mg_dose_placebo
- Normal_4mg Placebo: Normal_4mg_dose placebo
Arm/Group | Binge_4mg d | Normal_1mg d | Normal_2mg d | Normal_4mg d | Binge - 4mg Plc | Normal 1 mg Placebo | Normal 2mg_placebo | Normal_4mg Placebo
Number analyzed (Participants) | 7 | 4 | 4 | 8 | 7 | 4 | 4 | 8
mm | 144.14 (1.82) | 101 (9.74) | 128.75 (9.84) | 103.13 (17.22) | 117.57 (14.64) | 79.75 (24.29) | 131.25 (9.15) | 126 (5.2)
Statistical Analysis 1: Comparison: Binge_4mg d vs Normal_4mg d vs Binge - 4mg Plc vs Normal_4mg Placebo; Each group was compared separately in an overall ANOVA with all dose groups included. The results are presented for the groups which received 4 mg dose and instructions to eat normally (normal group) or to binge eat (binge group). The test is the interaction between drug and group i.e. drug effect difference (placebo minus drug) in fullness between the group instructed to binge and the group instructed to eat normally; Test type: Superiority or Other; p = .033, t-test, 2 sided — t-test after ANOVA with repeated measures on placebo minus drug (within groups) between binge and normal instructions (between groups); This was part of an overall ANOVA (SAS proc mixed) with all four groups (3 doses eat normally. 4 ng dose, binge eat) and the error term had 76 df; Mean Difference (Final Values) = 49.4, Standard Error of Mean 22.8

3. Secondary Outcome: Sickness Report
Description: Response to question "How sick do you feel" measured on a 150 mm line anchored by none at all (0 mm left end) and extremely (150 mm right end)
Time Frame: 25-30 min after drug or placebo
Measure: Mean (Standard Error); unit: mm
Arm/Group | Binge_4mg Drug | Normal_1mg Drug | Normal_2mg Drug | Normal_4mg Drug | Binge - 4mg Placebo | Normal 1 mg Dose Placebo | Normal_2 mg Dose Placebo | Normal_4 mg Dose Placebo
Number analyzed (Participants) | 7 | 4 | 4 | 8 | 7 | 4 | 4 | 8
mm | 94.57 (22.48) | 21 (14.58) | 10 (7.07) | 17.5 (9.64) | 61.14 (20.79) | 3 (1.35) | 10 (8.72) | 17.25 (8.43)
Statistical Analysis 1: Comparison: Binge - 4mg Placebo vs Normal_4 mg Dose Placebo; Tests the difference between drug and placebo for group = binge instructions; Test type: Superiority or Other; p < .014, ANOVA — p-value is based on ANOVA with all groups and conditions and is a planned comparison; Mean Difference (Final Values) = 33.4286, Standard Error of Mean 13.134 — df = 53. 26 Used proc GLMMIX in SAS 9.4

ADVERSE EVENTS:
Time Frame: Length of the study - 2 - 4 weeks
Description: There were no adverse events reported.
Groups:
- Normal: Normal control group
Arm/Group | Normal
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

LIMITATIONS AND CAVEATS:
No adverse events - Some subjects reported a "sick" feeling that was significantly different between drug and control, in the condition where they were instructed to binge eat. This is a subtle feeling without any other symptoms. It is not adverse.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The provider of the drug (not sponsor - since this was an investigator initiated protocol) needs to review the results before release. In this case there was a public presentation at a scientific meeting, and the abstract was published. However, before a full report can be released, the provider of the drug needs to review the report.